CLINICAL TRIAL: NCT04556097
Title: Implementation of the Care Ecosystem Training Model for Individuals With Dementia in a High-risk, Integrated Care Management
Acronym: CRESCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brent Forester, Chief, Division of Geriatric Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020P000880
Record Dates: First submitted 2020-06-17; First posted 2020-09-21 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Training (Experimental): Nurse care managers will be randomized to either early or delayed adapted Care Ecosystem training. The Early Training arm will be the first group to receive training and the first to have the opportunity to use the training in a clinical setting. We anticipate that each nurse care manager will manage 10 PWLD and we anticipate a 50% response rate/data availability, yielding 75 patients per arm.
  Interventions: Behavioral: Care Ecosystem
- Delayed Training (Active Comparator): The Delayed Training arm will be the second group of nurse care managers to receive training.
  Interventions: Behavioral: Care Ecosystem

INTERVENTIONS:
Behavioral: Care Ecosystem — The Care Ecosystem model uses a telephone-based intervention to support persons with dementia and their care partners, screening for common dementia-related problems and providing modular standardized support protocols and caregiver education. Specially trained health care navigators systematically identify needs and address health status, advance care planning, medication management and management of challenging behaviors. Health care navigators receive backup support from a nurse, social worker, dementia specialist, and pharmacist, and maintain close communication with the primary care provider of the persons with dementia.
  This Care Ecosystem model will be adapted to augment the dementia care provided by experienced Integrated Care Management Program nurse care managers engaged in the care of high-risk, high-cost patients in a large health system.

SUMMARY:
There is growing need for to provide high quality care for persons living with dementia (PLWD) and provide support for care partners in the primary care setting. The Care Ecosystem model is a telephone-based dementia care program that provides standardized, proactive, personalized, and scalable support and education for care partners. The Care Ecosystem model has demonstrated an improvement in patient quality of life, reduced unnecessary healthcare expenditures, and a decrease in care partner burden and depression.

In this pilot the investigators will assess the feasibility of implementing and measuring outcomes of an adapted Care Ecosystem training model for primary care nurse managers serving a diverse panel of PLWD and their care partners in primary care practices participating in the Mass General Brigham healthcare system's Integrated Care Management Program in Boston, MA. The study team will leverage the Mass General Brigham electronic medical record to determine the feasibility of collecting the primary clinical outcome defined as emergency department visits among the PLWD cared for by the primary care practices. The investigative team will also assess the feasibility of implementation, number of contacts between nurse care managers and care partners, and documented advance care planning.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiary aligned to the Partners Medicare ACO
* ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019 and July 31, 2020 (excluding diagnoses for diagnostic testing services)
* Actively engaged in care management services with a nurse care manager enrolled in the study

Exclusion Criteria:

- Permanent resident of long-term care or deceased at the start of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 524 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellinger TJ, Forester BP, Vogeli C, Donelan K, Gulla J, Vetter M, Vienneau M, Ritchie CS. Impact of dementia care training on nurse care managers' interactions with family caregivers. BMC Geriatr. 2023 Jan 11;23(1):16. doi: 10.1186/s12877-022-03717-w. PMID 36631767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a pragmatic trial where nurse managers at various primary care practices were randomized to the control group which had delayed training or the intervention group which was the early intervention training. The enrollment number in the protocol section conflicts with the number of participants started in the flow module as some patients without a designated caregiver, who were deceased or who had moved to a skilled nursing facility were excluded.
Groups:
- Intervention- PWD: Patients of nurse care managers who received adapted Care Ecosystem training in December 2020 and January 2021.
- Control- PWD: Patients of nurse care managers who did not receive adapted Care Ecosystem training in December 2020 and January 2021.
- Intervention - NCM: Nurse care managers who received adapted Care Ecosystem training in December 2020 and January 2021. Their patients are persons with dementia and their primary caregiver under the care of these nurse care managers were defines as Medicare beneficiaries aligned to the Mass General Brigham Medicare ACO with an ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019, and July 31, 2020.
- Control- NCM: Nurse care managers who did not receive adapted Care Ecosystem training in December 2020 and January 2021. Their patients are persons with dementia and their primary caregiver under the care of these nurse care managers were defines as Medicare beneficiaries aligned to the Mass General Brigham Medicare ACO with an ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019, and July 31, 2020.
Period: Overall Study
Arm/Group | Intervention- PWD | Control- PWD | Intervention - NCM | Control- NCM
Started | 206 | 187 | 15 | 15
Mailed Caregiver Survey | 143 | 113 | 0 (Nurse care managers did not complete the surveys.) | 0 (Nurse care managers did not complete the surveys.)
Completed Baseline Survey | 57 | 43 | 0 (Nurse care managers did not complete the surveys.) | 0 (Nurse care managers did not complete the surveys.)
Completed 6-month Follow-up Survey | 35 | 26 | 0 (Nurse care managers did not complete the surveys.) | 0 (Nurse care managers did not complete the surveys.)
Completed | 126 | 105 | 14 | 15
Not Completed | 80 | 82 | 1 | 0
Not completed — Death | 0 | 5 | 0 | 0
Not completed — No caregiver | 43 | 53 | 0 | 0
Not completed — Ineligible, SNF | 2 | 2 | 0 | 0
Not completed — Ineligible, health | 3 | 4 | 0 | 0
Not completed — Ineligible, language | 0 | 1 | 0 | 0
Not completed — Ineligible, no longer in care management | 0 | 2 | 1 | 0
Not completed — No dementia | 13 | 3 | 0 | 0
Not completed — Missing identifier | 2 | 4 | 0 | 0
Not completed — Did not have at least 1 member month in pre and post period | 17 | 8 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population for the primary outcome of Emergency Department visits was restricted to only include those PWD who had at least 1 member month during pre-intervention and post-intervention. The analysis population for the outcome of NPI-Q Distress among caregivers for persons with dementia was further restricted only to those who completed the baseline and 6-month follow-up surveys (Intervention, N=35; Control, N=28).
Groups:
- Intervention- PWD: Persons with Dementia Intervention: Patients of nurse care managers who received adapted Care Ecosystem training in December 2020 and January 2021.
- Control- PWD: Persons with Dementia Control: Patients of nurse care managers who did not receive adapted Care Ecosystem training in December 2020 and January 2021.
- Intervention- NCM: Nurse Care Managers Intervention: Nurse care managers who received adapted Care Ecosystem training in December 2020 and January 2021. Their patients are persons with dementia and their primary caregiver under the care of these nurse care managers were defines as Medicare beneficiaries aligned to the Mass General Brigham Medicare ACO with an ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019, and July 31, 2020.
- Control- NCM: Nurse Care Managers Control: Nurse care managers who did not receive adapted Care Ecosystem training in December 2020 and January 2021. Their patients are persons with dementia and their primary caregiver under the care of these nurse care managers were defines as Medicare beneficiaries aligned to the Mass General Brigham Medicare ACO with an ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019, and July 31, 2020.
- Total: Total of all reporting groups
Arm/Group | Intervention- PWD | Control- PWD | Intervention- NCM | Control- NCM | Total
Number analyzed (Participants) | 126 | 105 | 14 | 15 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 14 | 15 | 34
  >=65 years | 126 | 100 | 0 | 0 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not measured for nurse care managers in the intervention or control groups.
  years
    number analyzed (Participants) | 126 | 105 | 0 | 0 | 231
    (all) | 84.83 (8.17) | 82.88 (9.37) |  |  | 83.94 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 68 | 12 | 13 | 175
  Male | 44 | 37 | 2 | 2 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 6 | 0 | 0 | 25
  Not Hispanic or Latino | 103 | 97 | 0 | 0 | 200
  Unknown or Not Reported | 4 | 2 | 14 | 15 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 3 | 0 | 0 | 12
  White | 93 | 94 | 0 | 0 | 187
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 24 | 8 | 14 | 15 | 61
Region of Enrollment [Number; unit: participants]
  United States | 126 | 105 | 14 | 15 | 231
ED Visits Per Member Per Month [Mean (Standard Deviation); unit: Visits per member per month] — Count of emergency department visits within 6 months prior to the intervention based on Medicare parts A and B. Emergency department visits resulting in inpatient admission will be excluded. Population: Measure was not collected for nurse care managers as it only applies to PWD.
  Visits per member per month
    number analyzed (Participants) | 126 | 105 | 0 | 0 | 231
    (all) | 0.060 (0.158) | 0.052 (0.080) |  |  | 0.057 (0.128)
NPI-Q Distress Score [Mean (Standard Deviation); unit: Score on a scale] — The NPI-Q has 12 items assessing caregiver distress associated with dementia patient's behaviors. Participant distress is rated for each positive neuropsychiatric symptom domain on a scale anchored by score from 0 to 5 points. The Score is: 0 = Not distressing at all, 1 = Minimal (slightly distressing, not a problem to cope with), 2 = Mild (not very distressing, generally easy to cope with), 3 = Moderate (fairly distressing, not always easy to cope with), 4 = Severe (very distressing, difficult to cope with), 5 = Extreme of Very Severe (extremely distressing, unable to cope with) Population: The analysis population for the outcome of NPI-Q Distress among caregivers for persons with dementia was restricted only to those who completed the baseline and 6-month follow-up surveys (Intervention, N=35; Control, N=28). Measure was not collected for NCMs as it only applies to PWD.
  Score on a scale
    number analyzed (Participants) | 35 | 28 | 0 | 0 | 63
    (all) | 11.17 (9.27) | 9.29 (6.41) |  |  | 10.33 (8.12)

OUTCOME MEASURES:

1. Primary Outcome: ED Visits Per Member Per Month 6 Months Post Intervention
Time Frame: 6 months
Population: The analysis population for the primary outcome of Emergency Department visits includes all patients eligible for the baseline survey who had at least 1 member month during pre-intervention and post-intervention.
Measure: Mean (Standard Deviation); unit: Visits per member per month
Groups:
- Intervention: Persons with dementia and their primary caregiver who were under the care of nurse care managers who received adapted Care Ecosystem training in December 2020 and January 2021. Persons with dementia were defined as Medicare beneficiaries aligned to the Mass General Brigham Medicare ACO with an ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019 and July 31, 2020.
- Control: Persons with dementia and their primary caregiver who were under the care of nurse care managers who did not receive adapted Care Ecosystem training in December 2020 and January 2021. Persons with dementia were defined as Medicare beneficiaries aligned to the Mass General Brigham Medicare ACO with an ICD-10 diagnosis code consistent with dementia in Medicare claims between August 1, 2019 and July 31, 2020.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 126 | 105
Visits per member per month | 0.056 (0.129) | 0.075 (0.144)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.05, Difference in differences; Difference in differences model with a negative binomial distribution and log link that provides rate ratio estimate of the relative difference; Rate Ratio = 0.61, 95% CI 2-sided [0.31 to 1.20], Standard Error of Mean 0.35 — The rate ratio is estimated for intervention patients as compared to controls

2. Secondary Outcome: Caregiver Distress (NPI-Q) 6 Months Post
Description: Mean Neuropsychiatric Inventory Questionnaire (NPI-Q) distress score at 6-month follow-up survey. The NPI-Q distress scale assesses caregiver distress. Scores can range from 0 to 60 and higher scores indicate greater distress.
Time Frame: 6 months
Population: The analysis population for the outcome of NPI-Q Distress among caregivers for persons with dementia was restricted only to those who completed the baseline and 6-month follow-up surveys (Intervention, N=35; Control, N=28).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 35 | 28
Score on a scale | 10.86 (8.79) | 11.68 (8.60)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.05, Difference in differences; Difference in differences model with a Gaussian distribution and identity link that provides linear estimate of the relative point difference; Mean Difference (Net) = -2.7, 95% CI 2-sided [-6.53 to 1.12], Standard Error of Mean 1.95

ADVERSE EVENTS:
Time Frame: 6 months post period
Groups:
- Control-PWD: Persons with Dementia Control: Patients of nurse care managers who did not receive adapted Care Ecosystem training in December 2020 and January 2021.
Arm/Group | Intervention- PWD | Control-PWD | Intervention- NCM | Control- NCM
All-Cause Mortality (participants affected / at risk) | 21/126 | 14/105 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/105 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/126 | 0/105 | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04556097/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04556097/SAP_001.pdf